CLINICAL TRIAL: NCT05088499
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: The Role of Genetic Factors in the Development of Epilepsy in the Kazakh Population
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1199
Record Dates: First submitted 2021-09-25; First posted 2021-10-22 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy
Keywords: GWAS
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: Patients with epilepsy
  Interventions: Genetic: DNA analysis
- Control group: Patients without epilepsy
  Interventions: Genetic: DNA analysis

INTERVENTIONS:
Genetic: DNA analysis — GWAS

SUMMARY:
This is a GWAS study that aims to identify possible candidate genes associate to epilepsy by exploring single nucleotide polymorphism (SNP) in a group of epilepsy, in the Kazakh population. The investigators hypothesize that the careful phenotyping of the subject sand matching with increase the power to find SNP significantly associate with epilepsy

DETAILED DESCRIPTION:
A genome-wide association study (GWAS) is an approach used in genetics research to associate specific genetic variations with particular diseases. The method involves scanning the genomes from many different people and looking for genetic markers that can be used to predict the presence of a disease. Once such genetic markers are identified, they can be used to understand how genes contribute to the disease and develop better prevention and treatment strategies

ELIGIBILITY:
Inclusion Criteria:

* Children with seizures, confirmed by EEG and no morphological damage to the brain, confirmed by MRI of the brain;
* The age of the patients is from 0 to 5 years;
* Persons of Kazakh nationality, whose paternal and maternal grandparents are Kazakhs;
* Children are parents or legal guardians who have given written informed consent.

Exclusion Criteria:

* Children over 5 years old;
* Children whose parents, according to the researcher, are mentally or legally incapacitated, which prevents obtaining informed consent;
* Children with seizures with brain damage that cause epilepsy;
* Children of a non-Kazakh ethnic group.

Ages: 0 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: Children of Kazakh ethnic group
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
number of SNPs associated with epilepsy | 1 year
  Using GWAS to identify candidate genes associate with epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Altynshash Jaxybayeva, Study Director — Astana Medical University, Nur-Sultan, Kazakhstan
Locations (1):
- Altynshash Jaxybayeva, Almaty, Kazakhstan